CLINICAL TRIAL: NCT02138968
Title: Clinical and Economic Assessment of an Opportunistic Screening Program for Pre-frailty State in Elderly Population.
Brief Title: Clinical and Economic Assessment of a Pre-frail Screening Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17/13; CEIC 17/13 (Other: CEIC)
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pre-frail; Elderly
Keywords: Pre-frailty; Frail; Exercise; Nutritional assessment; Functional capacity
MeSH Terms: conditions — Motor Activity

ARMS (2):
- Multidimensional intervention (Experimental): Multidimensional intervention based on: good control of baseline diseases, review of medication adequacy, exercise program, nutritional assessment and control, social assessment and control.
  Interventions: Other: Multidisciplinary intervention
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Multidisciplinary intervention — Multidimensional intervention based on: good control of baseline diseases, review of medication adequacy, exercise program, nutritional assessment and control, social assessment and control.
  Arms: Multidimensional intervention

SUMMARY:
The study intervention improves functional capacity and delays frailty status in pre-frail elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* More than 70 years consulting in primary care
* Non institutionalized
* Pre-frailty according to L.Fried criteria (1 or 2 criteria)
* Signed informed consent

Exclusion Criteria:

* Patient not able to stand by himself/herself
* Dementia
* Palliative care or life expectancy less than 6 months
* Blind patient
* unstable clinical situation
* Participation in other programs, studies or trials for elderly people

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Frailty according to L.Fried criteria (questionnaire). | One year
  L.Fried frailty criteria: (Robust: 0 criteria; Pre-frail: 1-2 criteria; Frail: >=3 criteria)
  1. Weight loss
  2. Fatigue
  3. Poor physical activity
  4. Low walking speed
  5. Low muscle strength Reference of L.Fried: J Gerontol A Biol Sci Med Sci. 2001 Mar; 56(3):M146-56. PMID: 11253156.
Functional capacity according to Barthel score and Timed up and go test. | One year
  Barthel score and Timed up and go test.

SECONDARY OUTCOMES:
Nutritional status according to MNA-sf. | One year
  Mini Nutritional Assessment short form (MNA-sf).
Quality of live according to EuroQoL. | One year
  EuroQoL.
Mortality | One year
Health resource consumption (composite measure) | One year
  Number of visits to primary care center, number of visits to hospital emergency department, number of hospitalizations, days of hospital stay, institutionalization to nursing homes, visits to nutritionist and visits to social services.

OTHER OUTCOMES:
Pain according Visual Analog Scale. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mateu Serra-Prat, PhD, Principal Investigator — Fundació Salut del Consorci Sanitari del Maresme
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Serra-Prat M, Sist X, Domenich R, Jurado L, Saiz A, Roces A, Palomera E, Tarradelles M, Papiol M. Effectiveness of an intervention to prevent frailty in pre-frail community-dwelling older people consulting in primary care: a randomised controlled trial. Age Ageing. 2017 May 1;46(3):401-407. doi: 10.1093/ageing/afw242. PMID 28064172